CLINICAL TRIAL: NCT00467402
Title: A 52-week, Randomized, Double-blind, Placebo-controlled, Multi-center, Parallel-group Study of the Long-term Efficacy, Tolerability and Safety of Agomelatine 25 and 50 mg in the Prevention of Relapse of Major Depressive Disorder (MDD) Following Open-label Treatment of 16-24 Weeks
Brief Title: Efficacy, Safety and Tolerability of Agomelatine in the Prevention of Relapse of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAGO178A2304
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
Keywords: agomelatine, Major Depressive Disorder, MDD, depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: agomelatine
- 2 (Experimental)
  Interventions: Drug: agomelatine
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: agomelatine
  Arms: 1; 2
Drug: placebo
  Arms: 3

SUMMARY:
This study will demonstrate the efficacy of agomelatine (AGO178) 25 mg and 50 mg in the prevention of relapse in patients with Major Depressive Disorder (MDD). Eligible patients will undergo open-label treatment for 20 to 26 weeks, depending on response to treatment. Patients demonstrating stable response at the end of the open-label treatment phase will be assigned to receive agomelatine or placebo for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 through 70 years of age, inclusive
* Diagnosis of Major Depressive Disorder, recurrent episode, according to Diagnostic and Statistical Manual of Mental Disorders - 4th Edition (DSM-IV) criteria
* A history of at least two previous episodes of Major Depression plus the current episode
* Hamilton Depression Rating Scale (HAM-D17) total score ≥ 22 at Screening and Baseline

Exclusion Criteria:

* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder, or obsessive compulsive disorder
* Any current Axis I disorder other than major depressive disorder which is the focus of treatment
* Substance or alcohol abuse in the last 30 days, dependence in the last 6 months
* Use of any psychoactive medication after the screening visit
* Patients who have been previously treated with agomelatine
* Female patients of childbearing potential who are not using effective contraception

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Time to relapse, where relapse is defined by the occurrence of any one of the following: | Primary efficacy variable is measured from randomization to relapse
Hamilton Depression Rating Scale total score ≥16 at two consecutive visits; | Primary efficacy variable is measured from randomization to relapse
hospitalization due to depression; | Primary efficacy variable is measured from randomization to relapse
suicide attempt or suicide; | Primary efficacy variable is measured from randomization to relapse
discontinuation due to lack of efficacy according to Investigator judgment. | Primary efficacy variable is measured from randomization to relapse

SECONDARY OUTCOMES:
Proportion of patients who demonstrate clinical improvement at the end of the double-blind continuation phase, where improvement is defined by a score of 1 or 2 on the Clinical Global Impression Improvement (CGI-I) scale. | Secondary efficacy variables will be measured from randomization to the end of the Double-Blind continuation Phase
Proportion of patients experiencing relapse during the double-blind continuation phase. | Secondary efficacy variables will be measured from randomization to the end of the Double-Blind continuation Phase
Proportion of patients who achieve remission at the end of the double-blind continuation phase, where remission is defined by a total score of ≤7 on the HAM-D. | Secondary efficacy variables will be measured from randomization to the end of the Double-Blind continuation Phase
Change from randomization to the end of the double-blind continuation phase, on the Hospital Anxiety and Depression (HAD) total score and subscale scores. | Secondary efficacy variables will be measured from randomization to the end of the Double-Blind continuation Phase

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Costa Mesa, California
  - Novartis Investigative Site, Encino, California
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Sherman Oaks, California
  - Novartis Investigative Site, Temecula, California
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Coral Springs, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Venice, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Libertyville, Illinois
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Towson, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Braintree, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Farmington Hills, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Rhododendron, Oregon
  - Novartis Investigative Site, Allentown, Pennsylvania
  - Novartis Investigative Site, Lansdale, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, DeSoto, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lake Jackson, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Virginia Beach, Virginia
  - Novartis Investigative Site, Edmonds, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
  - Novartis Investigative Site, West Allis, Wisconsin

REFERENCES:
- See also: Results for CAGO178A2304 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3420